CLINICAL TRIAL: NCT02091934
Title: A Prospective, Randomized Comparison of Fellow Eyes Undergoing Wavefront-guided PRK Versus Wavefront-optimized PRK Using the Alcon Allegretto Eye-Q 400 Excimer Laser
Brief Title: Wavefront-guided PRK vs Wavefront-optimized PRK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Edward E. Manche, Professor of Ophthalmology, Stanford University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Stanford IRB #29233
Record Dates: First submitted 2014-03-09; First posted 2014-03-19 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Myopia; Astigmatism
Keywords: Alcon; Wavelight; PRK; Wavefront-guided; Wavefront-optimized; Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wavefront-guided PRK (Active Comparator): Wavefront-guided PRK
  Interventions: Procedure: Wavefront-guided PRK
- Wavefront-optimized PRK (Active Comparator): Wavefront-optimized PRK
  Interventions: Procedure: Wavefront-optimized PRK

INTERVENTIONS:
Procedure: Wavefront-guided PRK — Wavefront-guided PRK
  Other Names: Alcon Wavelight Eye-Q 400 wavefront-guided PRK
  Arms: Wavefront-guided PRK
Procedure: Wavefront-optimized PRK — Wavefront-optimized PRK
  Other Names: Alcon Wavelight Eye-Q 400 wavefront-optimized PRK
  Arms: Wavefront-optimized PRK

SUMMARY:
The purpose of the study is to compare the results of PRKK surgery when using wavefront-guided excimer laser treatment compared to wavefront optimized excimer laser treatment in patients with nearsightedness with and without astigmatism

DETAILED DESCRIPTION:
This is a research study comparing the outcomes of PRK surgery for nearsightedness when using the two different excimer laser technologies. Patients will have both eyes treated with the Alcon WaveLight Allegretto excimer laser. You will be one of 50 sighted patients at Stanford to undergo treatment in this clinical research trial. This will be a prospective, randomized, research study in which up to 100 consecutive eyes scheduled to undergo excimer laser photo refractive keratectomy (PRK) using one laser technology in the first eye and the second laser technology in the fellow eye for the correction of myopia (nearsightedness) with or without astigmatism will be enrolled. The choice of which eye receives the wavefront guided technology and which eye receives the wavefront-optimized technology will be randomized prior to enrollment. Randomization will be done according to a randomization schedule. You will not know which eye is being treated with which each technology. The randomization will determine only whether your right or left eye is treated with the wavefront guided technology. The other eye will be treated with wavefront-optimized laser technology. You have a fifty percent chance of having your left eye treated with custom wavefront guided technology as your right eye. Subjects will undergo bilateral (both eyes at once) PRK treatments using the Alcon WaveLight Allegretto excimer laser. All subjects will be followed for one year after the vision correction procedure. Subjects scheduled to undergo PRK for the correction of myopia (nearsightedness) with or without astigmatism will be screened for eligibility. Eligible subjects will be examined preoperatively to establish a baseline for ocular condition (the general health and glasses prescription of the eyes). Postoperatively, subjects will undergo an ophthalmic evaluation (complete eye examination) at regular intervals as specified in this protocol. Patients will complete questionnaires preoperatively and postoperatively evaluating quality of vision and quality of life. Retreatments (a second operation on the same eye for residual nearsightedness) will not be allowed during the first twelve months of this study. If you elect to undergo a retreatment of your PRK surgery prior to the 12-month post-operative visit, the retreated eye will be exited from the study as of the retreatment date.

Any significant new finding developed during the course of the research which may relate to the subject's willingness to continue participation will be provided to the subject or subject's representative in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 21 and older with healthy eyes.
* Nearsightedness between -0.25 diopters and -8.00 diopters with or without astigmatism of up to 5.00 diopters.

Exclusion Criteria:

* Subjects under the age of 21.
* Excessively thin corneas.
* Topographic evidence of keratoconus.
* Ectactic eye disorders.
* Autoimmune diseases.
* Pregnant or nursing.
* Patients must have similar levels of nearsightedness in each eye. They can not be more than 2.5 diopter of difference between eyes.
* Patients must have similar levels of astigmatism in each eye. They can not have more than 1.5 diopter of difference between eyes.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2009-04-01 (Actual); Primary Completion 2012-03-31 (Actual); Study Completion 2012-03-31 (Actual)

PRIMARY OUTCOMES:
Uncorrected visual acuity | One year
  Uncorrected visual acuity

SECONDARY OUTCOMES:
Topographic analysis | One year
  Topographic analysis
Wavefront analysis | One year
  Wavefront analysis
Quality of vision and quality of life questionnaire | One year
  Patient Reported Outcomes Questionnaire
Corneal haze | One year
  Corneal haze
Changes in best corrected 5 and 25% contrast visual acuity | One year
  Changes in best corrected 5 and 25% contrast visual acuity
Changes in best corrected visual acuity | One year
  Changes in best corrected visual acuity
Refractive predictability | One year
  Refractive predictability

CONTACTS AND LOCATIONS:
Overall Officials: Edward E Manche, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Eye Laser Center, Palo Alto, California, United States

REFERENCES:
- [Result] He L, Manche EE. Contralateral eye-to-eye comparison of wavefront-guided and wavefront-optimized photorefractive keratectomy: a randomized clinical trial. JAMA Ophthalmol. 2015 Jan;133(1):51-9. doi: 10.1001/jamaophthalmol.2014.3876. PMID 25321951